CLINICAL TRIAL: NCT04919993
Title: Cognitive Behavioral Therapy for Insomnia in Primary Brain Tumor Patients
Brief Title: CBT for Insomnia in Primary Brain Tumor Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-20-16188
Record Dates: First submitted 2021-05-24; First posted 2021-06-09 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Primary Brain Tumor; PBT
Keywords: Cognitive Behavioral Therapy-Insomnia; CBT-I
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase IIa Proof-of-Concept Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy for Insomnia (CBT-I) (Experimental): Group intervention; topics include psychoeducation about sleep, sleep restriction, stimulus control, relaxation strategies, and cognitive restructuring.
  Interventions: Behavioral: Cognitive Behavioral Therapy-Insomnia

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy-Insomnia — Group presentation
  Other Names: CBT-I

SUMMARY:
The purpose of this study is to pilot test an empirically supported psychotherapeutic intervention, Cognitive Behavior Therapy for Insomnia (CBT-I) in primary brain tumor patients. Researchers hope to better understand the feasibility and acceptability of this intervention in neuro-oncology, as well as the preliminary potential benefits of this intervention on brain tumor patients' sleep, fatigue, mood, quality of life, and chronic inflammation. This may lead to improvements in treating insomnia in primary brain tumor patients.

DETAILED DESCRIPTION:
The present study design is a pilot within-subjects pre-/post-evaluation of feasibility, acceptability, and preliminary efficacy of the Cognitive Behavioral Therapy for Insomnia (CBT-I) intervention for primary brain tumor patients. In this study, participants will be asked to do the following things:

* Meet with a trained interventionist six times (biweekly) for group CBT-I sessions via Zoom, lasting 90 minutes each. Participants will be asked to only use first names and will complete weekly sleep diaries as part of the intervention.
* Complete ~20-minute online surveys before the program, immediately after the program (6 weeks), and at follow-up (3 months). Questions will ask about subjective sleep, fatigue, mood, and quality of life. The follow-up time point will also ask about the patient's satisfaction with the CBT-I program.
* Complete a brief (15 minute) cognitive evaluation before and immediately following the program.
* Wear a wrist-worn actigraphy monitor one week prior to the 6-week CBT-I intervention and one week following completion of the intervention.
* Patients currently receiving regular blood draws as part of their care at Massey Cancer Center will have an IL-6 added to their regular blood draw. THose who are not receiving regular blood draws as part of their standard of care OR those who are not patients at Massey Cancer Center will forego this part of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years old
* Confirmed primary brain tumor diagnosis
* >/= 1 month removed from radiation therapy (if applicable)
* Able to readily read and understand English
* Meeting DSM-V diagnostic criteria for insomnia as measured by the Structured Clinical Interview for DSM-5
* Sleep Disorders (SCISD) insomnia subsection
* Cognitively intact as measured by a score >20 on the Telephone Interview for Cognitive Status (TICS)
* Have a stable internet connection and video-capable device for Zoom sessions

Exclusion Criteria:

* Inability to attend weekly group in-person meetings
* Patients must also meet the inclusion criteria listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Feasibility for CBT-I as measured by the rates of participant screening, eligibility, and consent | 12 months
  Determine how many patients consent to screening after referral to the program, how many patients are eligible for the program after being screened, and how many consent/enroll in the program if eligible.
Attendance at CBT-I sessions | 6 weeks
  Percent of sessions attended by consented participants
Post-session assessment completion | 2 months
  Percent of post-session surveys completed by participants immediately after the intervention
Follow-up assessment completion | 5 months
  Percent of follow-up surveys completed by participants three months after the intervention
Program Satisfaction as measured by participant responses to researcher-developed questions (e.g., How satisfied were you with the program overall?) measured on a Likert scale | 7 months
  Program satisfaction questions are measured on a 10-point Likert scale with 1 being not at all satisfied and 10 being very much satisfied. Higher scores indicate greater program satisfaction.

SECONDARY OUTCOMES:
Objective Sleep | 7 months
  Total sleep time gathered by the participant from a wrist-worn Actigraph
Sleep Efficiency | 7 months
  Percent of time spent in bed / time asleep gathered by the participant from a wrist-worn Actigraph
Subjective Sleep | 7 months
  Total sleep time gathered from a participant-reported sleep diary
Subjective Insomnia | 7 Months
  Determine the degree of participant insomnia using the Insomnia Severity Index, a brief self-report questionnaire measured on a 5-point Likert scale (0 = None, 4 = Very Severe). Higher scores indicate greater subjective insomnia.
Subjective Sleep Disturbance | 7 Months
  Determine the degree of participant sleep disturbance using the Pittsburgh Sleep Quality Index, a brief self-report questionnaire. Higher scores indicate greater global sleep disturbance.
Napping | 7 Months
  Request that participants self report how many hours a day they nap on average using one self-report question (During the past month, how many hours did you nap during a typical day?)
Fatigue | 7 Months
  Determine participants' level of fatigue using the Brief Fatigue Inventory, a self-report questionnaire measured on a 11-point Likert scale (0 = No Fatigue/Does Not Interfere; 10 = As Bad as You Can Imagine/Completely Interferes). Higher scores indicate greater symptoms of fatigue.
Depression | 7 Months
  Determine the extent of depressive symptoms using the Patient Health Questionnaire-9, a brief-self report questionnaire measured on a 4-point Likert scale (0 = Not at All; 3 = Nearly Everyday) Higher scores indicate greater symptoms of depression.
Anxiety | 7 Months
  Determine the extent of anxiety symptoms using the Generalized Anxiety Disorder-7, a self-report questionnaire measured on a 4-point Likert scale (0 = Not at All; 3 = Nearly Everyday). Higher scores indicate greater symptoms of anxiety.
Death Anxiety | 7 Months
  Determine the level of participant's death anxiety using the Death and Dying Distress Scale, a self-report questionnaire measured on a 6-point Likert scale (0 = Not Distress; 5 = Extreme Distress). Higher scores indicate greater symptoms of death anxiety.
Subjective Quality of Life as measured by participants' responses on the European Organization Research and Treatment of Cancer - Quality of Life - Cancer 30 (EORTC-QoL-C30) form. | 7 Months
  Determine participants' level of quality of life using the EORTC-QoL-C30, a self-report questionnaire measured on a 4-point Likert scale (1 = Not at All; 4 = Very Much). Higher scores indicate lower overall quality of life.
Inflammation | 7 Months
  Determine the level of inflammation as measured by the amount of Cytokine Interleukin-6 (IL-6) in the participant's blood; only participants receiving regular blood draws as part of their routine will have this data
Processing Speed | 7 months
  Participants' speed of thinking will be assessed by administering the Trail Making Test A, a neuropsychological assessment tool
Executive Function | 7 months
  Measure executive functioning by administering the Trail Making Test B, a neuropsychological assessment tool
Language Fluency | 7 months
  Participants' language fluency will be measured using the Controlled Oral Word Association Test, a neuropsychological assessment tool
Learning/Memory | 7 months
  Participants' ability learn/ memory will be assessed by administering the Hopkins Verbal Learning Test, a neuropsychological assessment tool
Sociodemographics | 7 months
  Participants are requested to self-report on their age, gender identity, race/ethnicity, and level of education
Primary Brain Tumor Characteristics | 7 months
  Information on participants' tumor diagnosis, treatment history, and medications will be from the participants' medical charts to determine brain tumor characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Ashlee Loughan, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan in place to share data with other researchers.

REFERENCES:
- [Derived] Loughan AR, Lanoye A, Willis KD, Fox A, Ravyts SG, Zukas A, Kim Y. Telehealth group Cognitive-Behavioral Therapy for Insomnia (CBT-I) in primary brain tumor: Primary outcomes from a single-arm phase II feasibility and proof-of-concept trial. Neuro Oncol. 2024 Mar 4;26(3):516-527. doi: 10.1093/neuonc/noad193. PMID 37796017

DOCUMENTS (1):
  • Informed Consent Form (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT04919993/ICF_002.pdf